CLINICAL TRIAL: NCT03605901
Title: Dosing of Methadone for Spine Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201700673; OCR18737 (Other: University of Florida)
Record Dates: First submitted 2018-07-18; First posted 2018-07-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative
Keywords: Post-operative pain; Spine surgery; Methadone; Opioid
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two different protocols by a designated study team member based on a computer generated randomization table. Randomization will occur on the day of surgery. Randomization will be 1:1.
Who Masked: Outcomes Assessor
Masking Description: Post-operative data will be collected by blinded staff. Patient daily pain based on the analog scale of 0-10 post-operative for the first 72 hours, total opioid usage, length of stay, time to get out of bed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dosing of methadone (Active Comparator): Receive 0.2 mg/kg based on ideal body weight of methadone after the intubation and before positioning.
  Interventions: Drug: Standard dosing of methadone
- Aliquots of methadone titrated to apnea (Experimental): Receive incremental aliquots of methadone up to 0.5 mg/Kg based on ideal body weight titrated to apnea. Each subject will receive a 5-10 mg loading dose then aliquots of 5mg each, given at 3 to 5 minute time intervals. The practitioner will continue to coach patient to take deep breaths. After reaching the apnea threshold as determined by respiratory rate less than 8 breaths/min, induction of general anesthesia and intubation will proceed.
  Interventions: Drug: Aliquots of methadone titrated to apnea

INTERVENTIONS:
Drug: Standard dosing of methadone — Subject will receive 0.2 mg/kg based on ideal body weight of methadone after the intubation and before positioning.
  Arms: Standard dosing of methadone
Drug: Aliquots of methadone titrated to apnea — Subjects will receive incremental aliquots of methadone up to 0.5 mg/Kg based on ideal body weight titrated to apnea. Each subject will receive a 5-10 mg loading dose then aliquots of 5mg each, given at 3 to 5 minute time intervals.
  Arms: Aliquots of methadone titrated to apnea

SUMMARY:
This study compares two methods of dosing methadone for complex spine cases

DETAILED DESCRIPTION:
Patients with spine surgery experience a significant amount of pain that can interfere with healing, rehabilitation and contribute to morbidity in the post-operative period. This study will compare post-operative opioid requirement at 24 and 48 hours to determine if methadone given in small aliquots until respiratory depression can act as a self-control to determine the correct dose required.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must consent to participate and sign the IRB-approved informed consent prior to beginning any study specific procedures.
2. At or between the ages 18 to 75 years.
3. Undergoing multilevel thoracic, thoracolumbar and/or lumbar spine surgery with instrumentation and fusion.

Exclusion Criteria:

1. Methadone or buprenorphine use.
2. Morbid obesity with BMI>40 Kg/m2.
3. Chronic renal failure with creatinine>2.0 mg/dL.
4. Liver failure as determined by cirrhosis or history of fulminant hepatic failure.
5. Current or historical alcohol abuse.
6. Current or historical drug abuse.
7. Patients with history of prolonged QTc, as defined as a QTc value >450 ms in males and >460 ms in females.
8. Patients with ASA status IV or V.
9. Surgical diagnosis including spine tumor, infection, or trauma.
10. In the Principal Investigator's opinion is not a candidate for the study.
11. Unwilling to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Change in opioid requirement for complex spine surgery patients | Changes from baseline (pre-op) up to 72 hours post-op
  Titrating methadone to respiratory depression allows the patient to act as his own control determining the dose he will require, improving pain control and consequently decreasing side effects and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Seubert, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538